CLINICAL TRIAL: NCT06667921
Title: The Diagnostic Efficacy of Ultrasonographic Airway Assessment in Predicting Difficult Laryngoscopy in Pediatric Patients Undergoing Elective Surgery; A Prospective Observational Study
Brief Title: Ultrasonographic Airway Assessment in Predicting Difficult Laryngoscopy in Pediatric Patients Undergoing Elective Surgery
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Mostafa El-Sayed Abo Farrag, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36265MD172/11/23
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Ultrasonographic; Airway; Difficult Laryngoscopy; Pediatric; Elective Surgery
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasonographic group: Ultrasound will be used to measure the hyomental distance in neutral position (HMDRn), hyomental distance in extended position (HMDRe), (HMDR) and (DSE).
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound will be used to measure the hyomental distance in neutral position (HMDRn), hyomental distance in extended position (HMDRe), (HMDR) and (DSE).

SUMMARY:
This study aims to evaluate the diagnostic accuracy of ultrasonographic airway examination in predicting difficult laryngoscopy in pediatric patients undergoing elective surgery.

DETAILED DESCRIPTION:
A difficult airway in a paediatric patient can be a stressful situation for anaesthesiologists as the most common causes of anaesthesia-related deaths were the result of difficult intubation, which is a more common problem in children than in adults.

Ultrasonography is a valuable, promising tool for preoperative airway evaluation through identifying important son anatomy of the upper airway, such as epiglottis, thyroid cartilage, and vocal cords.

Many studies have shown that some ultrasonic parameters can predict difficult airways in adults, such as tongue thickness, hyomental distance in the extended position (HMDE), distance from skin to epiglottis (DSE), tongue volume, midsagittal tongue cross-sectional area (TCSA), and tongue width. However, whether these parameters can be used to predict difficult laryngoscopy in children is unclear and needs extensive studies

ELIGIBILITY:
Inclusion Criteria:

* Children aged (2-5) years old.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I or II.
* Undergoing elective surgery under general anaesthesia with endotracheal intubation.

Exclusion Criteria:

* Maxillofacial trauma
* Large mass.
* Scar under the chin.
* History of neck surgery or congenital anomalies of the head and neck as difficult intubation is expected in these cases.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This prospective observational study will be carried out on 308 children of both genders, American Society of Anesthesiology (ASA) physical status I or II, who will be prepared for elective surgery under general anaesthesia with tracheal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of ultrasound measurement of hyomental distance ratio (HMDR) | 10 minutes till placement of endotracheal tube
  Accuracy of ultrasound measurement of hyomental distance ratio (HMDR) in predicting difficult laryngoscopy will be recorded

SECONDARY OUTCOMES:
Accuracy of ultrasound measurement of distance from skin to epiglottis (DSE) | 10 minutes till placement of endotracheal tube
  Accuracy of ultrasound measurement of distance from skin to epiglottis (DSE) in predicting difficult laryngoscopy
Correlation between the pre-anaesthetic ultrasonographic airway assessment, hyomental distance ratio (HMDR) and distance from skin to epiglottis (DSE) | 10 minutes till placement of endotracheal tube
  Correlation between the pre-anaesthetic ultrasonographic airway assessment, hyomental distance ratio (HMDR) and distance from skin to epiglottis (DSE), with the modified Cormack-Lehane grade of direct laryngoscopic view under general anaesthesia.
  The laryngoscopic view of the patient's airway will be graded using the Modified Cormack and Lehane grading scale; grades 1 and 2 are considered easy laryngoscopy, and grades 3 and 4 are considered difficult laryngoscopy.
  Grade 1: the whole glottis is visible. Grade 2: part of the cords is visible. Grade 3: only epiglottis is visible. Grade 4: epiglottis isn't visible.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.